CLINICAL TRIAL: NCT00702468
Title: A Placebo Controlled, Parallel Group, Randomised Withdrawal Study of Subjects With Symptoms of Spasticity Due to Multiple Sclerosis Who Are Receiving Long-term Sativex®.
Brief Title: Evaluate the Maintenance of Effect After Long-term Treatment With Sativex® in Subjects With Symptoms of Spasticity Due to Multiple Sclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: GWSP0702
Record Dates: First submitted 2008-06-19; First posted 2008-06-20 (Estimated); Results first posted 2011-06-17 (Estimated); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Spasticity; Multiple Sclerosis
Keywords: Spasticity; Multiple Sclerosis
MeSH Terms: conditions — Muscle Spasticity; Multiple Sclerosis | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sativex (Experimental): Sativex
  Interventions: Drug: Sativex
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sativex — containing delta-9-tetrahydrocannabinol (THC)(27 mg/ml):cannabidiol (CBD)(25 mg/ml), in ethanol:propylene glycol (50:50) excipients, with peppermint oil (0.05%) flavouring. Dose: 100 µl oromucosal spray, as required for symptom relief
  Other Names: GW-1000-02
  Arms: Sativex
Drug: Placebo — Contains no active drug and is delivered in 100 microlitre actuations by a pump action oromucosal spray
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the maintenance of effect after long-term treatment with Sativex® in subjects with symptoms of spasticity due to Multiple Sclerosis (MS) who have been receiving long-term benefit from treatment with Sativex®.

DETAILED DESCRIPTION:
This five week (one week baseline and four weeks randomised treatment period), multi-centre, placebo controlled, parallel group, randomized withdrawal study will evaluate the maintenance of effect after long-term treatment with Sativex® in subjects with symptoms of spasticity due to MS who have been receiving long-term benefit from treatment with Sativex®. Subjects will be selected from the Supply of Unlicensed Sativex® (SUS) or named patient supply programmes and must have been receiving Sativex® for at least 12 weeks prior to study entry. Following informed consent and screening, eligible subjects will enter the study (Visit 1, Day 1) and commence a seven day open label baseline period, before returning for a randomisation visit (Visit 2, Day 7), at which point they are randomised to receive either Sativex® or placebo (randomised withdrawal period). Subjects will return to the centre for an end of study visit at week five (Visit 3, Day 35) or earlier if they withdraw from treatment. Spasticity and sleep disruption review and dosing diaries will be completed each day from the start of the baseline period until completion or withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent for participation in the study.
* Male or female, aged 18 years or above.
* Subject is able (in the investigator's opinion) and willing to comply with all study requirements.
* Diagnosed with MS.
* Received Sativex for the relief of spasticity for at least 12 weeks prior to screening and willing to stop dosing with their own supply for the duration of the study.
* Judged to have been receiving benefit from and shown tolerability to Sativex, in the investigators' and subjects' opinion.
* Takes a minimum dose of Sativex of two sprays per day.
* If receiving disease-modifying medications, these must have been at a stable dose for at least three months prior to screening, and willing to maintain this for the duration of the study.
* Has had a stable regimen for at least 30 days prior to study entry, for all medications and non-pharmacological therapies that may have an affect on spasticity; and willing to maintain this for the duration of the study (N.B. This should be three months prior to study entry, in the case of Interferon therapy).
* Willing to allow his or her general practitioner and consultant, if appropriate, to be notified of participation in the study.
* Willing for his or her name to be notified to the responsible authorities for participation in this study

Exclusion Criteria:

* Has any concomitant disease or disorder that has symptoms of spasticity or that may influence the subject's level of spasticity.
* Unable to rate their level of spasticity or distinguish it from other MS symptoms.
* Currently receiving a prohibited medication (Botulinum Toxin, or Acomplia (Rimonabant), and unwilling to stop or comply for the duration of the study or had received said medication/ therapy within three months prior to the screening visit.
* Unwilling to stop their own Sativex treatment for the duration of the study.
* Any known or suspected immediate family history of schizophrenia, other psychotic illness, severe personality disorder or other significant psychiatric disorder other than depression associated with their underlying condition.
* Has evidence of cardiomyopathy.
* Has experienced myocardial infarction or clinically relevant cardiac dysfunction within the last 12 months or has a cardiac disorder that, in the opinion of the investigator would put the subject at risk of a clinically relevant arrhythmia or myocardial infarction.
* Has a QT interval of > 450 ms (males) or > 470 ms (females) at Visit 1.
* Has a secondary or tertiary atrioventricular (AV) block or sinus bradycardia (HR <50bpm unless physiological) or sinus tachycardia (HR>110bpm) at Visit 1.
* Has a diastolic blood pressure of <50 mmHg or >105 mmHg (when measured in a sitting position at rest for five minutes) prior to randomisation
* Has impaired renal function e.g. creatinine clearance is lower than 50ml/min at Visit 1 and is indicative of renal impairment.
* Has significantly impaired hepatic function, at Visit 1, in the investigator's opinion.
* Female subjects of child bearing potential and male subjects whose partner is of child bearing potential, unless willing to ensure that they or their partner use effective contraception during the study and for three months thereafter.
* Female subject who is pregnant, lactating or planning pregnancy during the course of the study and for three months thereafter.
* Subjects who have received any IMP within the 12 weeks before Visit 1.
* Any other significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, may influence the result of the study, or the subject's ability to participate in the study.
* Following a physical examination, the subject has any abnormalities that, in the opinion of the investigator, would prevent them from safely participating in the study.
* Travel outside the UK planned during the study.
* Unwilling to abstain from donation of blood during the study.
* Subjects previously randomised into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2007-11; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Notcutt, MB ChB, FRCA, Principal Investigator — James Paget University Hospital NHS Foundation Trust
Locations (1):
- James Paget University Hospital NHS Foundation Trust, Gorleston-on-Sea, Norfolk, United Kingdom

REFERENCES:
- [Result] Notcutt W, Langford R, Davies P, Ratcliffe S, Potts R. A placebo-controlled, parallel-group, randomized withdrawal study of subjects with symptoms of spasticity due to multiple sclerosis who are receiving long-term Sativex(R) (nabiximols). Mult Scler. 2012 Feb;18(2):219-28. doi: 10.1177/1352458511419700. Epub 2011 Aug 30. PMID 21878454
- [Derived] Di Marzo V, Centonze D. Placebo effects in a multiple sclerosis spasticity enriched clinical trial with the oromucosal cannabinoid spray (THC/CBD): dimension and possible causes. CNS Neurosci Ther. 2015 Mar;21(3):215-21. doi: 10.1111/cns.12358. Epub 2014 Dec 4. PMID 25475413

RESULTS

PARTICIPANT FLOW:
Groups:
- Sativex: Subjects received study medication delivered in 100 microlitre actuations by a pump action oromucosal spray. Maximum permitted dose of eight actuations in any three hour period and 48 actuations (delat9-tetrahydrocannabinol (THC)130 mg: 27 mg/ml: cannabidiol (CBD) 120 mg) in 24 hours.
- Placebo: Subjects received placebo delivered in 100 microlitre actuations by a pump action oromucosal spray. Maximum permitted dose of eight actuations in any three hour period and 48 actuations in 24 hours.
Period: Overall Study
Arm/Group | Sativex | Placebo
Started | 18 | 18
Completed | 15 | 2
Not Completed | 3 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sativex | Placebo | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (8.97) | 54.4 (10.42) | 57.1 (9.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 12 | 21
  Male | 9 | 6 | 15
Duration of Multiple Sclerosis (MS) [Mean (Standard Deviation); unit: years] | 17.84 (8.48) | 15.05 (10.07) | 16.44 (9.29)
Duration of Spasticity [Mean (Standard Deviation); unit: years] | 14.38 (9.90) | 11.01 (8.25) | 12.69 (9.14)
Expanded Disability Status Scale (EDSS) Score [Median (Full Range); unit: Score on scale] — The EDSS is an ordinal clinical rating scale ranging from 0 (normal neurologic examination) to 10 (death due to MS) in half-point increments.
  Score on scale | 7.0 (1.67) [4.0 to 8.5] | 7.0 (2.23) [5.5 to 8.5] | 7.0 (1.96) [4.0 to 8.5]
Baseline Spasticity Numerical Rating Scale (NRS) Score [Mean (Standard Deviation); unit: Score on scale] — Spasticity NRS was completed daily by answering the following question:
  "On a scale of '0 to 10' please indicate the average level of your spasticity over the last 24 hours" with the anchors: 0 = 'no spasticity' and 10 = 'worst possible spasticity'.
  Score on scale | 3.60 (1.67) | 4.13 (2.23) | 3.87 (1.96)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Experience Treatment Failure.
Description: The time to treatment failure was calculated as the number of days from the first day of treatment up to the day of treatment failure. The day of treatment failure was the earliest of:the day of premature cessation of study medication;the first day of the longest period, ending on the last day of treatment, where the mean spasticity NRS had increased by at least 20% and at least 1 unit from the treatment baseline; the day of a clinically relevant increase in anti-spasticity or disease modifying medication. The number of subjects who failed treatment were calculated.
Time Frame: Week 1- Week 5
Measure: Number; unit: Participants
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 18 | 18
Participants | 8 | 17
Statistical Analysis 1: Comparison: Sativex vs Placebo; Test type: Superiority or Other; p = 0.013, Chi-squared; Odds Ratio (OR) = 0.335, 90% CI 2-sided [0.162 to 0.691]

2. Secondary Outcome: Change in Mean Daily Spasticity Severity as Measured on a Spasticity Severity 0-10 Numerical Rating Scale (NRS).
Description: Spasticity NRS was completed daily by answering the following question:
  "On a scale of '0 to 10' please indicate the average level of your spasticity over the last 24 hours" with the anchors: 0 = 'no spasticity' and 10 = 'worst possible spasticity'. The change in mean spasticity severity NRS from baseline to end of study (last seven days)was calculated. A negative change from baseline indicates an improvement in spasticity.
Time Frame: Baseline (Week 1) to Week 5
Population: It is important to note that 17 of the placebo subjects withdrew from the study early. All subjects were accounted for in this analysis by use of a last-observation-carried-forward approach.
Measure: Mean (Standard Deviation); unit: points on scale
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 18 | 18
points on scale | 1.11 (1.92) | 1.10 (1.91)
Statistical Analysis 1: Comparison: Sativex vs Placebo; Test type: Superiority or Other; p = 0.720, ANCOVA; Estimated treatment difference = -0.21, 90% CI 2-sided [-1.22 to 0.79] — Negative difference indicates the comparison is in favour of Sativex

3. Secondary Outcome: Change in Modified Ashworth Scale.
Description: The Modified Ashworth Scale was completed at baseline and at the end of treatment at approximately the same time of day. All 20 muscle groups were assessed for spasticity (using a 0=no increase in muscle tone to 4 scale=affected part rigid in flexion or extensions), to result in a total score out of 80. The higher the score the worse the spasticity is.
  The change from baseline to end of study was assessed. The higher the score the better
Time Frame: Day 7 to Day 28
Population: ITT. The reason for not including some of the data in this analysis is that a number of the subjects who withdrew early from the study restarted their own Sativex before the assessment was done.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 17 | 8
score on scale | 21.5 (12.73) | 22.9 (17.11)
Statistical Analysis 1: Comparison: Sativex vs Placebo; Test type: Superiority or Other; p = 0.86, ANCOVA; Treatment difference = 0.53, 90% CI 2-sided [-4.68 to 5.74]

4. Secondary Outcome: Change in Motricity Index
Description: The Motricity Index involves assessing three movements in both the arms and the legs. In the arm the three movements are; pinch grip, elbow flexion and shoulder abduction and the three leg movements are, ankle dorsiflexion, knee extension and hip flexion. The total arm/leg score is then the addition of the score for the three arm/leg movements. One point is then added to each limb score so that the maximum score is 100 points. The higher the score the better the limb movement.
Time Frame: Week 2 and Week 5
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: points on scale
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 16 | 7
points on scale
  Arm | 72.4 (6.26) | 92.5 (0)
  Leg | 43.6 (31.40) | 47.0 (21.38)

5. Secondary Outcome: Timed 10-metre Walk.
Description: The time taken to travel 10 metres.
Time Frame: Week 2 and Week 5
Population: ITT. Only 4 placebo subjects were included in the analysis and 11 of the Sativex subjects. The reason for not including some of the data in this analysis is that a number of the subjects who withdrew early from the study restarted their own Sativex before the assessment was done.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 11 | 4
Seconds | 47.3 (50.29) | 18.3 (4.5)
Statistical Analysis 1: Comparison: Sativex vs Placebo; It is important to emphasise that only four placebo subjects were included in the analysis and 11 of the Sativex subjects - this sample size is too small for a meaningful comparison between treatments. The reason for not including some of the data in this analysis is that a number of the subjects who withdrew early from the study restarted their own Sativex before the assessment was done; Test type: Superiority or Other; p = 0.81, ANCOVA; Slope = -1.78, 90% CI 2-sided [-14.52 to 10.96] — Negative difference indicates the comparison is in favour of Sativex

6. Secondary Outcome: Daily Sleep Disruption NRS
Description: Subjects will be asked: "On a scale of 0-10 please indicate how your spasticity disrupted your sleep last night" with the anchors 0 = 'did not disrupt sleep', 10 = 'completely disrupted (unable to sleep at all)'.
Time Frame: Week 1- Week 5
Population: It is important to note that 16 of the placebo subjects withdrew from the study early. All subjects were accounted for in this analysis by use of a last-observation-carried-forward approach.
Measure: Mean (Standard Deviation); unit: points on scale
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 18 | 18
points on scale | 2.90 (2.48) | 3.36 (2.18)
Statistical Analysis 1: Comparison: Sativex vs Placebo; Test type: Superiority or Other; p = 0.271, ANCOVA; treatment difference = -0.64, 90% CI 2-sided [-1.60 to 0.33] — A negative difference indicates the comparison is in favour of Sativex

7. Secondary Outcome: Subject Global Impressions of Change.
Description: At baseline subjects will write a brief description of their spasticity caused by MS and how it affects them emotionally, physically and their ability to function with day to day activities. This will be used to aid their memory before they answer the following question which is rated on a seven-point scale.
  "Please assess the change in your spasticity due to MS since immediately before receiving the first course of study treatment (Baseline) using the scale below" The markers are: Very much worse, Much worse, Minimally worse, No change, Minimally better, Much better, Very much better.
Time Frame: Day 35
Measure: Number; unit: participants
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 18 | 18
participants
  Very much better | 0 | 0
  Much better | 0 | 0
  Minimally better | 0 | 0
  No change | 6 | 1
  Minimally worse | 6 | 5
  Much worse | 5 | 9
  Very much worse | 1 | 3
Statistical Analysis 1: Comparison: Sativex vs Placebo; Test type: Superiority or Other; p = 0.017, Regression, Logistic; Odds Ratio (OR) = 4.562, 90% CI 2-sided [1.585 to 13.997]

8. Secondary Outcome: Carer Global Impressions of Change for Functional Ability
Description: The main carer will be asked to assess the change in the subject's condition at the end of the study (completion or withdrawal). It consists of 2 question which is rated on a seven-point scale: Very much worse, Much worse, Minimally worse, No change, Minimally better, Much better, Very much better. The carer will be asked since visit 2 (baseline):
  "How has the subject's general functional abilities changed?" "How has the subject's ease of transfer?" Not all subjects had carers; a total of 18 subjects from each treatment, of which 10 from Sativex and 14 from placebo completed it.
Time Frame: Day 35
Measure: Number; unit: paticipants
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 10 | 14
paticipants
  Very Much Better | 0 | 0
  Much Better | 0 | 0
  Minimally Better | 0 | 0
  No Change | 3 | 0
  Minimally Worse | 5 | 3
  Much Worse | 2 | 9
  Very Much Worse | 0 | 2
Statistical Analysis 1: Comparison: Sativex vs Placebo; Test type: Superiority or Other; p = 0.0011, Regression, Logistic; Odds Ratio (OR) = 18.550, 90% CI 2-sided [3.942 to 118.773]

9. Secondary Outcome: Carer Global Impressions of Change for Ease of Transfer
Description: as for outcome 8
Time Frame: Day 35
Measure: Number; unit: paticipants
Arm/Group | Sativex | Placebo
Number analyzed (Participants) | 10 | 14
paticipants
  Very Much Better | 0 | 0
  Much Better | 0 | 0
  Minimally Better | 0 | 0
  No Change | 3 | 2
  Minimally Worse | 5 | 5
  Much Worse | 2 | 6
  Very Much Worse | 0 | 1
Statistical Analysis 1: Comparison: Sativex vs Placebo; Test type: Superiority or Other; p = 0.1151, Regression, Logistic; Odds Ratio (OR) = 3.444, 90% CI 2-sided [0.948 to 13.718]

ADVERSE EVENTS:
Time Frame: All AEs occurring from the time of consent to post study follow up (Visit 3) i.e. 5 weeks were collected. All deaths and SAEs occurring within 28 days of the final dose of sudy medication were also collected.
Description: All AEs occurring during the study were reported in the running logs at the back of the study case report form.
Arm/Group | Sativex | Placebo
Serious Adverse Events (participants affected / at risk) | 1/18 | 0/18
Other Adverse Events (participants affected / at risk) | 15/18 | 14/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sativex (N=18) | Placebo (N=18)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sativex (N=18) | Placebo (N=18)
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Mouth Ulceration (Gastrointestinal disorders) | 1 | 0
Stomach Discomfort (Gastrointestinal disorders) | 1 | 0
Vomitting (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 2 | 0
Pain (General disorders) | 2 | 7
Application site pain (General disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Gait disturbance (General disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 3 | 0
Cystitis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1
Oral Herpes (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Gamma-glutamyltransferase increase (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasticity (Nervous system disorders) | 2 | 3
Dizziness (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Multiple Sclerosis (Nervous system disorders) | 1 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Trigeminal neuralgia (Nervous system disorders) | 0 | 2
Depressed mood (Psychiatric disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Hypertonic Bladder (Renal and urinary disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Skin tightness (Skin and subcutaneous tissue disorders) | 0 | 1
Hot flush (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GW will coordinate the dissemination of data from this study and may solicit input and assistance from the principal investigator. All publications for example, manuscripts, abstracts, oral/slide presentations or book chapters based on this study, must be submitted to GW for corporate review before release.